CLINICAL TRIAL: NCT05157464
Title: Losartan Use to Mitigate Arthrofibrosis Following Total Join Arthroplasty
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was not initiated, no participants enrolled.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-00823
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Arthrofibrosis
Keywords: Total Knee Arthroplasty (TKA)
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled, open label, parallel two-arm design, single-center study to compare the use of losartan in the prevention of stiffness following total knee arthroplasty.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Losartan Group (Experimental)
  Interventions: Drug: Losartan
- Control Group (No Intervention): No additional steps in management are required for the control arm of the study.

INTERVENTIONS:
Drug: Losartan — Patients in this group will receive Losartan 12.5mg orally twice daily beginning 2 weeks preoperatively and continuing for 4 weeks postoperatively. Losartan is an Angiotensin II Receptor Blocker currently used in the treatment of hypertension.
  Arms: Losartan Group

SUMMARY:
Recent research has focused on methods to mitigate scar tissue formation and arthrofibrosis following surgery in hopes that patients may attain maximal range of motion goals, avoid manipulation and secondary surgery (i.e. revision arthroplasty), and improve their function. The synovial fluid milieu has also highlighted the role of local biochemical markers that may be implicated in the development of arthrofibrosis. Losartan is an angiotensin receptor blocker with inhibitory effects on transforming growth factor beta (TGF-b), largely implicated in tissue repair and fibrosis by way of SMAD protein signaling suppression, and has been used in orthopaedic sports medicine to prevent stiffness following hip arthroscopy. To date, this has not commonly been used at NYU Langone in orthopedic surgery. The purpose of this study is to evaluate the efficacy of losartan use pre- and post-operatively on range of motion and the incidence of manipulation under anesthesia following total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are candidates for elective primary total knee arthroplasty for a diagnosis of osteoarthritis or inflammatory arthritis.
2. Patients ≥18 years of age
3. Patients have been medically cleared and scheduled for surgery
4. Patients' primary care physician has verified that the patient can safely take the described dose of Losartan for the duration of the study period.

Exclusion Criteria:

1. Any contraindications to Losartan
2. Revision surgery
3. Surgery for fracture, infection, or malignancy
4. Patients with a diagnosis of post-traumatic arthritis
5. Bilateral, simultaneous surgery
6. Patients already taking an ACE-inhibitor or Angiotensin receptor blocker for hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-Operative Range of Motion (ROM) | 90 days post-surgery
  ROM will be reported as the degree of knee flexion.
Post-Operative Rate of Manipulation under Anesthesia (MUA) | 90 days post-surgery
  Rate of MUA will be reported as percentage of participants that require MUA.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Rozell, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access upon reasonable request. Requests should be directed to daniel.waren@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.